CLINICAL TRIAL: NCT03484572
Title: Prevalence of Undernutrition in Assiut University Children Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereny Merzik, principle investigator, Assiut University
Other Study IDs: Prev U
Record Dates: First submitted 2018-03-24; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Undernutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Anthropometric measures — Weight (kg),Height (cm)Body mass index(kg/m²),Mid-upper arm-circumference(cm), tricipital skinfold (cm)

SUMMARY:
To describe the prevalence of undernutrition in infants and children admitted to Assiut university children hospital and to describe risk group and decrease length of stay in hospital.

DETAILED DESCRIPTION:
Malnutrition is defined as a state in which a deficiency (or excess) of energy, protein, and other nutrition causes measurable adverse effects on the body and on growth (in children), and may impact clinical outcome. Recent studies in developed countries have estimated the prevalence of malnutrition in hospitalized children as 12% to 24%. Causes of malnutrition: There are many types of malnutrition, and they have different causes. Some causes include: Poor diet, Starvation due to food not being available , Eating disorders, Problems with digesting food or absorbing nutrients from food , Certain medical conditions that make a person unable to eat Malnourished children were classified according to the type of malnutrition into: Acute malnutrition (wasting) , Chronic malnutrition (stunting) , Micronutrient malnutrition. Malnourished children experience more complications, such as infections after surgery, than well-nourished children, also leading to increased length of stay. In infants, early malnutrition is associated with delayed physical as well as intellectual development.

ELIGIBILITY:
Inclusion Criteria:

* All infants and children from 2 months to 6 years admitted to Assiut university children hospital .

Exclusion Criteria:

* Infants less than month ,Children over the age of 6 years .

Ages: 1 Month to 6 Years | Sex: All
Age Groups: Child
Study Population: Anthropometric measures will be done to all infants and children from 2months to 6 years who admitted to Assiut university children hospital by fulfilling check lists on admission and on discharge include weight,height,body mass index,mid upper arm circumference,tricipital fold.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Describe the prevalence of undernutrition in all infants and children admitted to Assiut university children hospital | Baseline
  Analysis of the prevalence of undernutrition (undernutrition rate) among pediatric patients at the time of hospital admission throughout a calendar year in Assiut university children hospital and identify types of undernutrition among those pediatric patients.

REFERENCES:
- [Background] Freijer K, van Puffelen E, Joosten KF, Hulst JM, Koopmanschap MA. The costs of disease related malnutrition in hospitalized children. Clin Nutr ESPEN. 2018 Feb;23:228-233. doi: 10.1016/j.clnesp.2017.09.009. Epub 2017 Oct 13. PMID 29460804
- [Background] Groleau V, Thibault M, Doyon M, Brochu EE, Roy CC, Babakissa C. Malnutrition in hospitalized children: prevalence, impact, and management. Can J Diet Pract Res. 2014 Spring;75(1):29-34. doi: 10.3148/75.1.2014.29. PMID 24606957
- [Background] Aurangzeb B, Whitten KE, Harrison B, Mitchell M, Kepreotes H, Sidler M, Lemberg DA, Day AS. Prevalence of malnutrition and risk of under-nutrition in hospitalized children. Clin Nutr. 2012 Feb;31(1):35-40. doi: 10.1016/j.clnu.2011.08.011. Epub 2011 Sep 25. PMID 21945311
- [Background] Joosten KF, Hulst JM. Prevalence of malnutrition in pediatric hospital patients. Curr Opin Pediatr. 2008 Oct;20(5):590-6. doi: 10.1097/MOP.0b013e32830c6ede. PMID 18781124
- [Background] Pawellek I, Dokoupil K, Koletzko B. Prevalence of malnutrition in paediatric hospital patients. Clin Nutr. 2008 Feb;27(1):72-6. doi: 10.1016/j.clnu.2007.11.001. Epub 2007 Dec 20. PMID 18086508
- [Background] Joosten KF, Hulst JM. Malnutrition in pediatric hospital patients: current issues. Nutrition. 2011 Feb;27(2):133-7. doi: 10.1016/j.nut.2010.06.001. Epub 2010 Aug 13. PMID 20708380
- [Background] Campanozzi A, Russo M, Catucci A, Rutigliano I, Canestrino G, Giardino I, Romondia A, Pettoello-Mantovani M. Hospital-acquired malnutrition in children with mild clinical conditions. Nutrition. 2009 May;25(5):540-7. doi: 10.1016/j.nut.2008.11.026. Epub 2009 Feb 20. PMID 19230617